CLINICAL TRIAL: NCT05997030
Title: Early Feasibility Study of Low-Intensity Focused Ultrasound (LIFU) Neuromodulation in Patients With Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease
Brief Title: Low-Intensity Focused Ultrasound (LIFU) Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, Director RNI, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RNI_NMD_AD01
Record Dates: First submitted 2023-08-04; First posted 2023-08-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neuromodulation (Experimental): Subjects meeting eligibility criteria will undergo Exablate low intensity focused ultrasound neuromodulation
  Interventions: Device: low intensity focused ultrasound (LIFU)

INTERVENTIONS:
Device: low intensity focused ultrasound (LIFU) — Subjects will undergo undergo a single LIFU of the target brain region

SUMMARY:
This study is a prospective, single-center, single-arm early feasibility study, to establish safety and tolerability of LIFU for neuromodulation in patients with mild cognitive impairment ( MCI) due to Alzheimer's disease.

DETAILED DESCRIPTION:
The primary objective is to evaluate the safety, feasibility and tolerability of LIFU as an adjunct neuromodulatory treatment for MCI due to AD

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females, aged 45-85 years
* Able and willing to give informed consent
* Must meet the clinical criteria for MCI due to Alzheimer's disease
* If receiving concurrent treatment with an AChEI and/or memantine, has been on a stable dose for at least 45 days
* Able to communicate sensations during the LIFU procedure

Exclusion Criteria:

* Unable to undergo MR-imaging because of implanted pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent make-up or small metal fragments in the eye that welders and other metal workers may have, or if candidates are uncomfortable in small spaces (have claustrophobia).
* Participants with more than 30% of the skull area traversed by the sonication pathway are covered by scars, scalp disorders (e.g., eczema), atrophy of the scalp, or implanted objects in the skull or the brain.
* Participants with a history of seizure disorder.
* Participants with clinically significant chronic pulmonary disorders e.g., severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area.
* Participant does not speak English
* Participant is pregnant or planning to be pregnant

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment Emergent Adverse Events | baseline and 7 and days after study procedure
  Safety will be assessed by recording all adverse events that are treatment related. Each Adverse Event will be documented for patterns of occurence.
Cognitive Change | baseline and 7 days after procedure
  Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)

SECONDARY OUTCOMES:
Imaging Changes | baseline, 7 and 30 days
  Changes in brain metabolism and connectivity using PET and fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, Principal Investigator — WVU Rockefeller Neuroscience Institute
Locations (1):
- Rockefeller Neuroscience Institute at West Virginia University, Morgantown, West Virginia, United States